CLINICAL TRIAL: NCT00853177
Title: MEOPA Breathing Analgesia vs Local Anesthesia for Oocyte Retrieval in ART: a Prospective, Randomized Controlled Study
Brief Title: MEOPA Breathing Analgesia for Oocyte Retrieval(KALOVAL)
Acronym: KALOVAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070304
Record Dates: First submitted 2009-02-06; First posted 2009-03-02 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2011-05

CONDITIONS: Infertility; Pain
Keywords: Oocyte retrieval; pain; surgery; anaesthesiology; Assisted Reproductive Technologies
MeSH Terms: conditions — Infertility; Pain | interventions — Lidocaine; Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nitrous oxide (Experimental): N2O of 50% and 50% O2
  MEOPA
  Interventions: Procedure: MEOPA inhalation
- lidocaine (Active Comparator): Injection solution 1%
  Interventions: Procedure: xylocaine

INTERVENTIONS:
Procedure: MEOPA inhalation — N2O of 50% and 50% O2
  Arms: nitrous oxide
Procedure: xylocaine — Ampoule-bottle of 20 ml
  Other Names: local anesthesia
  Arms: lidocaine

SUMMARY:
The purpose of this study is to assess pain, at or after oocyte retrieval, the effectiveness of self-controlled inhalation analgesia by nitrous oxide (N2O of 50% and 50% O2) by the patient compared to a local anesthesia combined with a tablet of 0.5 mg of Alprazolam.

DETAILED DESCRIPTION:
Oocyte retrieval is a major event during in VITRO-fertilization, with or without sperm micro-injection. Initially done by laparoscopy with general anesthesia, the oocyte collection is now carried out by trans-vaginal controlled ultrasound puncture. This potential painful event, related to trans-vaginal puncture or mechanical movements of the stimulated ovary, requires analgesia or anesthesia. General anesthesia is certainly effective in terms of collected oocytes. It remains, however, a heavy time consumer, with personal risks and distributor of anesthetic agents in blood or follicular fluid. These products could have a deleterious effect on early embryonic development or implantation. Few data are available concerning these risks in the literature. General anesthesia is still essential for pusillanimous patients or for patients with a heavy surgical past. Nitrous oxide is an inhaled gas with properties widely used in obstetric during parturition. It is regularly used during general anesthesia performed for oocyte retrieval. With a gas composed of 50% N2O and 50% O2, its main interest is to provide analgesia in a state of conscious sedation. The effects of nitrous oxide in this form had never been assessed on the clinical or biological Oocyte collection. We conducted a preliminary study to assess pain in patients receiving local anesthesia, according the current protocol. Thus, 44% of patients had severe pain (VAS> 40/100) during or just after transvaginal oocyte retrieval. In our preliminary experience, immediate or distance post-operative pain was high and we plan to evaluate the benefit of analgesia with nitrous oxide in terms of immediate post-operative pain with a prospective, randomized and controlled study as compared with local anesthesia associated to Alprazolam.

ELIGIBILITY:
Inclusion Criteria:

* patient requiring a first or second oocyte retrieval procedure for IVR or ICSI after ovarian stimulation by gonadotrophin
* agreement to participate to this study

Exclusion Criteria:

* absolute indication for oocyte retrieval with general anesthesia
* no agreement to participate to this study,
* painfully known patient-not easy ovarian vaginal accessibility for monitoring or puncture
* respiratory pathology-chronic liver, kidney pathology, immunodeficiency, -contraindication to the medications used during the protocol

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pain after oocyte retrieval at + 30, 60 and 120 minutes. | immediate (at + 30, 60 and 120 minutes)

SECONDARY OUTCOMES:
Patients satisfaction at time + 120 minutes. | immediate (at + 120 minutes)
Patients recommendation at time + 120 minutes. Patients with supplementary analgesics at time + 120 minutes. | immediate (at time + 120 minutes)
Patients with canceled protocol arm attribution during oocyte retrievalART already stated issues Reactive Oxygen Species in retrieved follicular fluid. | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Poncelet, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Jean Verdier, service de la médecine de la reproduction, avenue du 14 juillet, Bondy, Île-de-France Region, France

REFERENCES:
- [Result] Bauer C, Lahjibi-Paulet H, Somme D, Onody P, Saint Jean O, Gisselbrecht M. Tolerability of an equimolar mix of nitrous oxide and oxygen during painful procedures in very elderly patients. Drugs Aging. 2007;24(6):501-7. doi: 10.2165/00002512-200724060-00006. PMID 17571915
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pubmed/17571915?ordinalpos=2&itool=Entrez